CLINICAL TRIAL: NCT05376176
Title: A Phase IIa, Randomized, Double-Masked, Placebo-Controlled, Parallel-Group, Multicenter Study Assessing the Efficacy and Safety of STN1010904 Ophthalmic Suspension 0.03% and 0.1% Compared With Vehicle in Subjects With Fuchs Endothelial Corneal Dystrophy (FECD) - PHANTOM Study
Brief Title: A Multicenter Study Assessing the Efficacy and Safety of STN1010904 Ophthalmic Suspension 0.03% and 0.1% Compared With Vehicle in Subjects With Fuchs Endothelial Corneal Dystrophy (FECD)
Acronym: PHANTOM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Santen Inc. (Industry)
Collaborators: ActualEyes Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 101090401IN
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Fuchs Endothelial Corneal Dystrophy
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy | interventions — BID protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- STN1010904 ophthalmic suspension 0.03% BID (Experimental)
  Interventions: Drug: STN1010904 ophthalmic suspension 0.03% BID
- STN1010904 ophthalmic suspension 0.1% BID (Experimental)
  Interventions: Drug: STN1010904 ophthalmic suspension 0.1% BID
- Placebo Vehicle BID (Placebo Comparator)
  Interventions: Drug: Placebo (Vehicle) BID

INTERVENTIONS:
Drug: STN1010904 ophthalmic suspension 0.03% BID — 0.03% STN1010904 ophthalmic suspension BID
  Arms: STN1010904 ophthalmic suspension 0.03% BID
Drug: STN1010904 ophthalmic suspension 0.1% BID — 0.1% STN1010904 ophthalmic suspension BID
  Arms: STN1010904 ophthalmic suspension 0.1% BID
Drug: Placebo (Vehicle) BID — Placebo (vehicle) BID
  Arms: Placebo Vehicle BID

SUMMARY:
This is a Phase IIa study to assess efficacy and safety of STN1010904 ophthalmic suspension (0.03%, and 0.1 %), twice daily dosing when compared to Placebo in subjects diagnosed with Fuchs Endothelial Corneal Dystrophy (FECD). This study will consist of a Screening Period of up to 15 days and an 18-month Double-Masked Treatment Period, including 9 individual visits to the study site.

ELIGIBILITY:
Inclusion Criteria:

* Male or female diagnosed with FECD.

Exclusion Criteria:

* Females who are pregnant or lactating.
* Any ocular surgery for FECD (e.g., penetrating keratoplasty (PKP), Descemet stripping endothelial keratoplasty (DSEK), Descemet membrane endothelial keratoplasty (DMEK), Descemet stripping automated endothelial keratoplasty (DSAEK), Descemet stripping only (DSO) in the study eye.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2025-05-26 (Actual); Study Completion 2025-05-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline in best corrected visual acuity (BCVA) with contrast level of 100% at Month 18 | at 18 month
Change from baseline in BCVA with contrast level of 10% at Month 18 | at 18 month
Change from baseline in contrast sensitivity with glare light at Month 18 | at 18 month

SECONDARY OUTCOMES:
Best corrected visual acuity (BCVA) with contrast level of 100% at all post-baseline visits | up to month 18
BCVA with contrast level of 10% at all post-baseline visits | up to month 18
Contrast sensitivity with glare light at all post-baseline visits | up to month 18
Contrast sensitivity without glare light at all post-baseline visits | up to month 18

CONTACTS AND LOCATIONS:
Locations (15):
- United States (11):
  - Stein Eye Institution UCLA, Los Angeles, California
  - Price Vision Group, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Tauber Eye Center, Kansas City, Missouri
  - Comprehensive Eye Care, Ltd, Washington, Missouri
  - Metropolitan Eye Research and Surgery Center, Palisades Park, New Jersey
  - Devers Eye Institute, Portland, Oregon
  - Scott Christie and Associates, Cranberry Township, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - Houston Eye Associates, Houston, Texas
- France (2):
  - Fondation Ophtalmologique Adolphe de Rothschild, Paris
  - University Hospital of Saint-Etienne, Saint-Etienne
- India (2):
  - Medical Research Foundation, Chennai, Tamil Nadu
  - Suven Clinical Research CenterL V Prasad Eye Institute, Banjara Hills, Telangana